CLINICAL TRIAL: NCT03719391
Title: A Randomized, Open-Label, Cross-Over Study to Assess Nicotine Uptake and Subjective Measures With Use of JUUL 5% Electronic Nicotine Delivery Systems (ENDS) Compared to Usual Brand Combustible Cigarettes, a Comparator E-Cigarette, and Nicotine Gum in Healthy Adult Smokers
Brief Title: United States Pre-Market Tobacco Application Pharmacokinetics
Acronym: US-PMTA-PK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Juul Labs, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: PROT-00009
Record Dates: First submitted 2018-10-17; First posted 2018-10-25 (Actual); Last update posted 2021-06-14 (Actual); Status verified 2019-01

CONDITIONS: Nicotine Dependence; Nicotine Dependence, Cigarettes; Tobacco Use; Tobacco Smoking
Keywords: Electronic Nicotine Delivery System; Combustible Cigarettes; Nicotine
MeSH Terms: conditions — Tobacco Use Disorder; Tobacco Use; Tobacco Smoking; Vaping | interventions — Nicotine Chewing Gum

STUDY DESIGN:
Intervention Model Description: Randomized, Open-Label, Cross-Over
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (7):
- JUUL 5% Virginia Tobacco ENDS (Experimental): Treatment with JUUL Virginia Tobacco flavored 5.0% ENDS product.
  Interventions: Other: Virginia Tobacco flavored JUUL 5% ENDS
- JUUL 5% Cool Mint ENDS (Experimental): Treatment with JUUL Cool Mint flavored 5.0% ENDS product.
  Interventions: Other: Cool Mint flavored JUUL 5% ENDS
- JUUL 5% Mango ENDS (Experimental): Treatment with JUUL Mango flavored 5.0% ENDS product.
  Interventions: Other: Mango flavored JUUL 5% ENDS
- JUUL 5% Creme Brulee ENDS (Experimental): Treatment with JUUL Creme Brulee flavored 5.0% ENDS product.
  Interventions: Other: Creme Brulee flavored JUUL 5% ENDS
- VUSE Solo e-cigarette (Active Comparator): Treatment with VUSE Solo Original with 4.8% nicotine product.
  Interventions: Other: VUSE Solo e-cigarette
- Nicotine Gum (Active Comparator): Treatment with nicorette white ice mint 4mg nicotine polacrilex gum product.
  Interventions: Other: Nicorette White Ice Mint 4mg nicotine polacrilex gum
- Usual Brand Combustible Cigarette (Active Comparator): Treatment with usual brand combustible cigarette.
  Interventions: Other: Usual Brand combustible cigarette

INTERVENTIONS:
Other: Virginia Tobacco flavored JUUL 5% ENDS — Treatment with Virginia Tobacco flavored JUUL 5% ENDS (10 puffs).
  Other Names: JUUL
  Arms: JUUL 5% Virginia Tobacco ENDS
Other: Cool Mint flavored JUUL 5% ENDS — Treatment with Cool Mint flavored JUUL 5% ENDS (10 puffs).
  Other Names: JUUL
  Arms: JUUL 5% Cool Mint ENDS
Other: Mango flavored JUUL 5% ENDS — Treatment with Mango flavored JUUL 5% ENDS (10 puffs).
  Other Names: JUUL
  Arms: JUUL 5% Mango ENDS
Other: Creme Brulee flavored JUUL 5% ENDS — Treatment with Creme Brulee flavored JUUL 5% ENDS (10 puffs).
  Other Names: JUUL
  Arms: JUUL 5% Creme Brulee ENDS
Other: VUSE Solo e-cigarette — Treatment with VUSE Solo Original with 4.8% nicotine e-cigarette (10 puffs).
  Other Names: VUSE
  Arms: VUSE Solo e-cigarette
Other: Nicorette White Ice Mint 4mg nicotine polacrilex gum — Treatment with Nicorette White Ice Mint 4mg Nicotine polacrilex gum (30 minutes Chew and Park method)
  Other Names: Nicotine Gum
  Arms: Nicotine Gum
Other: Usual Brand combustible cigarette — Treatment with usual brand cigarette (10 puffs).
  Arms: Usual Brand Combustible Cigarette

SUMMARY:
A Randomized, Open-Label, Cross-Over Study to Assess Nicotine Uptake and Subjective Measures with Use of JUUL 5% Electronic Nicotine Delivery Systems (ENDS) Compared to Usual Brand Combustible Cigarettes, a Comparator E-Cigarette, and Nicotine Gum in Healthy Adult Smokers

DETAILED DESCRIPTION:
E-cigarettes may be an acceptable alternative to traditional cigarette smoking. In utilizing vaporization rather than combustion, the generation and inhaltion of smoke and carbon monoxide (CO) may be reduced or avoided. JUUL has developed several nicotine based liquid blends for use in e-cigarettes. This study will assess nicotine uptake during a 10-puff controlled and a 5-minute ad libitum use of four JUUL 5% electronic nicotine delivery systems (ENDS) relative to usual brand (UB) combustible cigarettes, a comparator electronic cigarette (e-cigarette), and nicotine gum.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, adult, male or female smoker, 21 to 65 years of age, inclusive
* Has been a smoker for at least 12 months prior to Screening. Brief periods of non-smoking (e.g., up to ~7 consecutive days due to illness, trying to quit, participation in a study where smoking was prohibited) during that time will be permitted at the discretion of the PI.
* Currently smokes an average of 10 or more king size or 100s manufactured combustible CPD, as reported at Screening.
* Has a positive urine cotinine (≥ 500 ng/mL) at Screening
* Has an exhaled CO > 12 ppm at Screening.
* Is willing to comply with the requirements of the study, including a willingness to use the study products during the study.

Exclusion Criteria:

* Has a history or presence of clinically significant gastrointestinal, renal, hepatic, neurologic, hematologic, endocrine, oncologic, urologic, pulmonary, immunologic, psychiatric, or cardiovascular disease, or any other condition that, in the opinion of the PI, would jeopardize the safety of the subject or impact the validity of the study results.
* Has a clinically significant abnormal finding on the physical examination, medical history, vital signs, ECG, or clinical laboratory results, in the opinion of the PI.
* Has a positive test for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg), or hepatitis C virus (HCV) at Screening.
* Has had an acute illness (e.g., upper respiratory infection, viral infection) requiring treatment within 14 days prior to Check-in.
* Has a fever (> 100.5°F) at Screening or Check-in.
* Has a body mass index (BMI) > 40.0 kg/m2 or < 18.0 kg/m2 at Screening.
* Has a history of drug or alcohol abuse within 24 months of Check-in, as determined by the PI.
* Has diabetes mellitus, asthma, or chronic obstructive pulmonary disease.
* Has a systolic blood pressure < 90 mmHg or > 150 mmHg, diastolic blood pressure < 40 mmHg or > 95 mmHg, or heart rate < 40 bpm or > 99 bpm at Screening.
* Has experienced an allergic reaction following previous e-cigarette use or with exposure to any primary components of the e-liquids (benzoic acid, propylene glycol and glycerol).
* Has an estimated creatinine clearance < 80 mL/minute (using the Cockcroft-Gault equation) at Screening.
* Has a positive urine screen for alcohol or drugs of abuse at Screening or Check-in.
* Has used medications known to interact with cytochrome P450 (CYP) 2A6 (including, but not limited to, amiodarone, amlodipine, amobarbital, buprenorphine, clofibrate, clotrimazole, desipramine, disulfiram, entacapone, fenofibrate, isoniazid, ketoconazole, letrozole, methimazole, methoxsalen, metyrapone, miconazole, modafinil, orphenadrine, pentobarbital, phenobarbital, pilocarpine, primidone, propoxyphene, quinidine, rifampicin, rifampin, secobarbital, selegiline, sulconazole, tioconazole, tranylcypromine) within 14 days or 5 half-lives of the drug, whichever is longer, prior to Check-in.
* Has used nicotine-containing products other than manufactured cigarettes (e.g., ENDS, roll-your-own cigarettes, bidis, snuff, nicotine inhaler, pipe, cigar, chewing tobacco, nicotine patch, nicotine spray, nicotine lozenge, or nicotine gum) within 14 days prior to Check-in.
* Has a prior history of JUUL product use prior to Screening
* Has used any prescription smoking cessation treatments, including, but not limited to, varenicline (Chantix®) or buproprion (Zyban®) within 3 months prior to Check-in.
* Is a self-reported puffer (i.e., adult smokers who draw smoke from the cigarette into the mouth and throat but do not inhale).
* Is planning to quit smoking during the study or postponing a quit attempt in order to participate in the study.
* Has donated plasma within 7 days prior to Check-in.
* Has donated blood or blood products (with the exception of plasma as noted above), had significant blood loss, or received whole blood or a blood product transfusion within 56 days prior to Check-in.
* Has participated in a previous clinical study for an investigational drug, device, biologic, or tobacco product within 30 days prior to Check-in.
* Is or has a first-degree relative (i.e., parent, sibling, child) who is a current employee of the study site.
* Is or has a first-degree relative (i.e., parent, sibling, child) who is a current employee, shareholder, or is member of the board of directors of JUUL Labs Inc.
* Has previously been diagnosed with any form of cancer, except for basal cell or squamous epithelial carcinomas of the skin that have been resected at least 1 year prior to Screening.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2018-10-19 (Actual); Primary Completion 2018-11-21 (Actual); Study Completion 2018-11-28 (Actual)

PRIMARY OUTCOMES:
To assess nicotine uptake during a 10-puff controlled use of four JUUL 5% electronic nicotine delivery systems (ENDS) relative to usual brand (UB) combustible cigarettes, a comparator electronic cigarette (e-cigarette), and nicotine gum. | 7 days
  Nicotine PK parameters will be calculated from the individual plasma concentrations per details provided in the SAP. Baseline adjustments to the (non-adjusted) PK endpoints will also be presented.

SECONDARY OUTCOMES:
To assess exhaled carbon monoxide [CO] following controlled use of four JUUL 5% ENDS relative to UB combustible cigarettes, a comparator e-cigarette, and nicotine gum | 7 Days
  Exhaled CO levels will be measured using a Bedfont Micro+ Smokerlyzer or similar device and levels at Screening and after product use will be assessed.
To assess measures of subjective effects with controlled use of four JUUL 5% ENDS relative to UB combustible cigarettes, a comparator e-cigarette, and nicotine gum using the "modified Product Evaluation Scale (mPES)" | 7 Days
  Change in Evaluation; Scale: 1 = not at all, 2 = very little, 3 = a little, 4 = moderately, 5 = a lot, 6 = quite a lot, 7 = extremely
  Four multi-item subscales will be derived from "Satisfaction" (items 1, 2, 3, and 12); "Psychological Reward" (items 4 through 8); "Aversion" (items 9, 10, 16, and 18); and "Relief" (item 11, 13, 14, 15, and reversed for item 19) and single items 17 and 20 will be summarized.
To assess blood pressure following controlled use of four JUUL 5% ENDS relative to UB combustible cigarettes, a comparator e-cigarette, and nicotine gum. | 7 Days
To assess heart rate following controlled use of four JUUL 5% ENDS relative to UB combustible cigarettes, a comparator e-cigarette, and nicotine gum. | 7 Days
To assess the safety and tolerability of short-term use of four JUUL 5% ENDS. | 7 Days
  Number of participants with Adverse Events associated with use of JUUL 5% Device will be described by individual listings and frequency tables.
To characterize product use of four JUUL 5% ENDS during controlled use sessions. | 7 Days
  All product use data will be summarized using descriptive statistics. The difference in weight pre- and post- product use of each JUUL product and comparator e-cigarettes will be summarized.
To assess measures of subjective effects with controlled use of four JUUL 5% ENDS relative to UB combustible cigarettes, a comparator e-cigarette, and nicotine gum using Intent to Use Again Questionnaire. | 7 Days
  The Intent to Use Again questionnaire will be assessed using a 100 mm bipolar VAS
To assess measures of subjective effects with controlled use of four JUUL 5% ENDS relative to UB combustible cigarettes, a comparator e-cigarette, and nicotine gum using Nicotine Withdrawal Questionnaire. | 7 Days
  The nicotine withdrawal will be assessed using a 100mm visual analog scale (VAS)
To assess measures of subjective effects with controlled use of four JUUL 5% ENDS relative to UB combustible cigarettes, a comparator e-cigarette, and nicotine gum using Product Direct Effect Questionnaire. | 7 Days
  Product direct effect will be assessed using a 100 mm VAS
To assess measures of subjective effects with controlled use of four JUUL 5% ENDS relative to UB combustible cigarettes, a comparator e-cigarette, and nicotine gum using Product Liking Questionnaire. | 7 Days
  Product liking will be assessed using a 100 mm VAS

CONTACTS AND LOCATIONS:
Locations (1):
- Vince & Associates Clinical Research, Overland Park, Kansas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jensen RP, Luo W, Pankow JF, Strongin RM, Peyton DH. Hidden formaldehyde in e-cigarette aerosols. N Engl J Med. 2015 Jan 22;372(4):392-4. doi: 10.1056/NEJMc1413069. No abstract available. PMID 25607446
- [Background] D'Ruiz CD, Graff DW, Robinson E. Reductions in biomarkers of exposure, impacts on smoking urge and assessment of product use and tolerability in adult smokers following partial or complete substitution of cigarettes with electronic cigarettes. BMC Public Health. 2016 Jul 11;16:543. doi: 10.1186/s12889-016-3236-1. PMID 27401980
- [Background] McNeill A et al. E-cigarettes: An Evidence Update. A report commissioned by Public Health England. Available at: https://www.gov.uk/government/uploads/system/uploads/ attachment_data/file/457102/Ecigarettes_an_evidence_update_A_report_commissioned_by_ Public_Health_England_FINAL.pdf (Aug 2015).
- [Background] Polosa R, Morjaria J, Caponnetto P, Caruso M, Strano S, Battaglia E, Russo C. Effect of smoking abstinence and reduction in asthmatic smokers switching to electronic cigarettes: evidence for harm reversal. Int J Environ Res Public Health. 2014 May 8;11(5):4965-77. doi: 10.3390/ijerph110504965. PMID 24814944
- [Background] Fagerstrom K. Determinants of tobacco use and renaming the FTND to the Fagerstrom Test for Cigarette Dependence. Nicotine Tob Res. 2012 Jan;14(1):75-8. doi: 10.1093/ntr/ntr137. Epub 2011 Oct 24. No abstract available. PMID 22025545
- [Background] Hatsukami DK, Zhang Y, O'Connor RJ, Severson HH. Subjective responses to oral tobacco products: scale validation. Nicotine Tob Res. 2013 Jul;15(7):1259-64. doi: 10.1093/ntr/nts265. Epub 2012 Dec 13. PMID 23239843
- [Background] HIPAA Privacy Rule. Information for Researchers. De-identifying Protected Health Information Under the Privacy Rule. U.S. Department of Health and Human Services. NIH (Feb 2007). Available at: http://privacyruleandresearch.nih.gov/pr_08.asp#8a. Last accessed 31-Jul-2017.